CLINICAL TRIAL: NCT03775213
Title: The Mathematics of Breast Cancer Overtreatment: Improving Treatment Choice Through Effective Communication of Personalized Cancer Risk
Brief Title: Acceptability of Active Monitoring (AM) as a Treatment Option for Ductal Carcinoma in Situ (DCIS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pro00101109; 4R00CA207872-03 (NIH)
Record Dates: First submitted 2018-12-11; First posted 2018-12-13 (Actual); Results first posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Ductal Carcinoma in Situ
Keywords: Ductal carcinoma in situ; Decision support tool; Informed decision-making; Overtreatment; Active surveillance; Active monitoring
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Treatment Options + Active Monitoring (Experimental): Participants explore decision support tool that includes current standard treatment options for DCIS, as well as active monitoring.
  Interventions: Behavioral: Decision Support Tool with Active Monitoring
- Standard Treatment Options (Active Comparator): Participants explore decision support tool that includes current standard treatment options for DCIS.
  Interventions: Behavioral: Decision Support Tool without Active Monitoring

INTERVENTIONS:
Behavioral: Decision Support Tool with Active Monitoring — The decision support tool communicates trade-offs for different management strategies for DCIS, including active monitoring and surgery options.
  Arms: Standard Treatment Options + Active Monitoring
Behavioral: Decision Support Tool without Active Monitoring — The decision support tool communicates trade-offs for different management strategies for DCIS, including surgery options only.
  Arms: Standard Treatment Options

SUMMARY:
The purpose of this research study is to evaluate a decision support tool for patients diagnosed with ductal carcinoma in situ (DCIS).

DETAILED DESCRIPTION:
Today, guideline concordant care options for patients diagnosed with ductal carcinoma in situ (DCIS) are lumpectomy (with or without radiation treatment) and mastectomy, with optional endocrine therapy. Several ongoing trials are evaluating the safety of active monitoring (AM) as an alternative to immediate surgery for select patient groups. Little is known about women's acceptability of AM after a diagnosis with DCIS.

Here the study team seeks to answer the question: if AM is found to be a safe alternative to immediate surgery, how likely are women to choose it as their first course of treatment?

In this study, women are asked to imagine having recently been diagnosed with DCIS. For some in the intervention arm, in-depth information about surgical options and AM are presented with a web-based decision support tool. After exploring the decision support tool, participants are asked to make a hypothetical treatment choice and to answer a series of additional questions about their decision-making process and personal preferences. Women in the control arm receive a reduced version of the decision support tool that only provides in-depth information about the surgical options (AM is mentioned as an experimental approach).

The overarching hypothesis of this study is that patients who are offered AM as a guideline-concordant care option (a potential future scenario if ongoing trials confirm the safety of AM) are more likely to choose it compared to women in current clinical practice (who receive information about surgical options only).

Primary research question: Compared to presenting active monitoring (AM) as an experimental option, does presenting AM as a guideline-concordant care option increase its uptake as treatment choice?

Secondary research questions: Compared to presenting active monitoring (AM) as an experimental option, does presenting active monitoring as a guideline-concordant care option increase AM acceptability, decrease perceived AM riskiness, and decrease uptake of mastectomy as treatment choice?

ELIGIBILITY:
Inclusion Criteria:

* Sex: Female
* Age: 50-79 years
* Has had a negative mammographic screen in the past 12 months

Exclusion Criteria:

* Personal history of breast cancer

Ages: 50 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc D Ryser, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Mammography Clinic, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Duke mammography clinics between October 2021 and January 2022. The first participant was enrolled on October 12th, 2021 and the last participant was enrolled on January 29th, 2022.
Groups:
- Standard Treatment Options + Active Monitoring (AM): Participants explore decision support tool that includes current standard treatment options for ductal carcinoma in situ (DCIS), as well as active monitoring (AM).
  Decision Support Tool with Active Monitoring: The decision support tool communicates trade-offs for different management strategies for DCIS, including active monitoring and surgery options.
- Standard Treatment Options: Participants explore decision support tool that includes current standard treatment options for ductal carcinoma in situ (DCIS).
  Decision Support Tool without Active Monitoring: The decision support tool communicates trade-offs for different management strategies for DCIS, including surgery options only.
Period: Overall Study
Arm/Group | Standard Treatment Options + Active Monitoring (AM) | Standard Treatment Options
Started | 160 | 162
Completed | 102 | 102
Not Completed | 58 | 60
Not completed — Withdrawal by Subject | 51 | 53
Not completed — Incomplete Survey | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Treatment Options + Active Monitoring | Standard Treatment Options | Total
Number analyzed (Participants) | 102 | 102 | 204
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64 [57 to 69] | 62 [56 to 67] | 62 [57 to 68]
Age, Customized [Count of Participants; unit: Participants]
  50-64 years | 55 | 61 | 116
  65-79 years | 47 | 41 | 88
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 102 | 204
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 69 | 63 | 132
  Black | 29 | 37 | 66
  Other | 4 | 2 | 6
Marital Status [Count of Participants; unit: Participants]
  In Relationship | 6 | 8 | 14
  Married | 73 | 60 | 133
  Divorced | 8 | 13 | 21
  Separated | 0 | 2 | 2
  Single | 14 | 15 | 29
  Other | 1 | 4 | 5
Education [Count of Participants; unit: Participants]
  Some High School | 2 | 1 | 3
  High School | 14 | 19 | 33
  Bachelor's Degree | 47 | 40 | 87
  Master's Degree | 29 | 30 | 59
  Professional Degree (e.g., MD, JD) | 5 | 9 | 14
  Doctorate Degree (e.g., PhD) | 5 | 3 | 8
Household Finances [Count of Participants; unit: Participants]
  Extra for special | 78 | 72 | 150
  Just enough | 16 | 23 | 39
  Cut back to pay bills | 8 | 3 | 11
  Difficulty paying bills | 0 | 4 | 4
Self-Reported Health Status, Median (Q1, Q3) [Median (Inter-Quartile Range); unit: units on a scale] — Self-Reported Health Status measured on a visual analog scale (0-100%), with 0 being the worst outcome and 100 being the best outcome.
  units on a scale | 83 [75 to 90] | 85 [75 to 90] | 83.5 [75 to 90]
Personal Cancer History [Count of Participants; unit: Participants] | 29 | 25 | 54
Family Cancer History [Count of Participants; unit: Participants] | 86 | 81 | 167
Maximizer Minimizer Scale, Median (Q1, Q3) [Median (Inter-Quartile Range); unit: units on a scale] — This categorical 6-point Likert scale ranges from "I strongly lean toward waiting and seeing" (1) to "I strongly lean toward taking action" (6). The scale captures the extent to which individuals are "medical maximizers" who are predisposed to seek health care even for minor problems, versus "medical minimizers" who prefer to avoid medical intervention unless it is necessary.
  units on a scale | 4.0 [2.0 to 5.0] | 4.0 [3.0 to 5.0] | 4.0 [2.5 to 5.0]
Graph Literacy Score (0-3), Median (Q1, Q3) [Median (Inter-Quartile Range); unit: units on a scale] — Single score derived from 3 items, each scored as correct or incorrect. Correct answers are summed for a total "graph literacy score" (0-3). Lower scores indicate worse outcomes, and higher scores indicate better outcomes.
  units on a scale | 2.0 [2.0 to 3.0] | 2.0 [2.0 to 3.0] | 2.0 [2.0 to 3.0]
Pre-tool Knowledge (1-5): Breast Cancer [Median (Inter-Quartile Range); unit: units on a scale] — 5-point Likert scale from "I know very little about breast cancer" (1) to "I know a lot about breast cancer" (5).
  units on a scale | 3.0 [2.0 to 3.0] | 3.0 [2.0 to 3.0] | 3.0 [2.0 to 3.0]
Pre-tool Knowledge (1-5): DCIS [Median (Inter-Quartile Range); unit: units on a scale] — 5-point Likert scale from "I know very little about DCIS" (1) to "I know a lot about DCIS" (5).
  units on a scale | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Chose Active Monitoring (AM).
Description: Presented to participants as a categorical item: active monitoring (AM), lumpectomy, lumpectomy with radiation, mastectomy. Recorded for analysis as binary: AM vs non-AM.
Time Frame: Up to 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Treatment Options + Active Monitoring | Standard Treatment Options
Number analyzed (Participants) | 102 | 102
Participants | 28 | 18
Statistical Analysis 1: Comparison: Standard Treatment Options + Active Monitoring vs Standard Treatment Options; Test type: Superiority; Risk Ratio (RR) = 1.53, 95% CI 2-sided [.91 to 2.58]

2. Secondary Outcome: Number of Participants Who Found the Treatment Option Acceptable.
Description: Acceptability was ascertained using 1-5 Likert scale. Acceptability, asked in terms of comfort with a given treatment choice, was anchored at 1="Not at all comfortable" and 5="Very comfortable." The outcome was dichotomized using responses of 4 or 5 to represent "Acceptable".
Time Frame: Up to 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Treatment Options + Active Monitoring | Standard Treatment Options
Number analyzed (Participants) | 102 | 102
Participants
  Active Monitoring | 32 | 32
  Lumpectomy | 50 | 47
  Lumpectomy with Radiation | 34 | 38
  Mastectomy | 18 | 22
Statistical Analysis 1: Comparison: Standard Treatment Options + Active Monitoring vs Standard Treatment Options; Active Monitoring; Test type: Superiority; Risk Ratio (RR) = .97, 95% CI 2-sided [.49 to 1.88]
Statistical Analysis 2: Comparison: Standard Treatment Options + Active Monitoring vs Standard Treatment Options; Lumpectomy; Test type: Superiority; Risk Ratio (RR) = 1.06, 95% CI 2-sided [.79 to 1.41]
Statistical Analysis 3: Comparison: Standard Treatment Options + Active Monitoring vs Standard Treatment Options; Lumpectomy with Radiation; Test type: Superiority; Risk Ratio (RR) = .90, 95% CI 2-sided [.62 to 1.30]
Statistical Analysis 4: Comparison: Standard Treatment Options + Active Monitoring vs Standard Treatment Options; Mastectomy; Test type: Superiority; Risk Ratio (RR) = .84, 95% CI 2-sided [.48 to 1.47]

3. Secondary Outcome: Number of Participants Who Perceived Active Monitoring as Risky.
Description: Perceived risk outcome was ascertained using 1-5 Likert scale. Perceived risk was asked for active monitoring only, and was anchored at 1="Not at all risky" and 5="Very risky". The outcome was dichotomized using responses of 4 or 5 to represent "Risky".
Time Frame: Up to 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Treatment Options + Active Monitoring | Standard Treatment Options
Number analyzed (Participants) | 102 | 102
Participants | 18 | 17
Statistical Analysis 1: Comparison: Standard Treatment Options + Active Monitoring vs Standard Treatment Options; Test type: Superiority; Risk Ratio (RR) = 1.08, 95% CI 2-sided [.59 to 1.98]

4. Secondary Outcome: Number of Participants Who Chose Mastectomy.
Description: Presented to participants as a categorical item: active monitoring, lumpectomy, lumpectomy with radiation, mastectomy. Recorded for analysis as binary: mastectomy vs non-mastectomy.
Time Frame: Up to 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Treatment Options + Active Monitoring | Standard Treatment Options
Number analyzed (Participants) | 102 | 102
Participants | 14 | 15
Statistical Analysis 1: Comparison: Standard Treatment Options + Active Monitoring vs Standard Treatment Options; Test type: Superiority; Risk Ratio (RR) = .96, 95% CI 2-sided [.65 to 1.45]

5. Secondary Outcome: Change in Self-perceived Knowledge About DCIS.
Description: Measured pre- and post-tool as a categorical 5-point Likert scale from "I know very little about DCIS" (1) to "I know a lot about DCIS" (5); analyzed as continuous variable.
Time Frame: Baseline and 1 hour
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Standard Treatment Options + Active Monitoring | Standard Treatment Options
Number analyzed (Participants) | 102 | 102
Units on a scale | 2 [2 to 3] | 2.5 [2 to 3]
Statistical Analysis 1: Comparison: Standard Treatment Options + Active Monitoring vs Standard Treatment Options; Test type: Superiority; Slope = .09, 95% CI 2-sided [-.20 to .38]

6. Other Pre Specified Outcome: Self-reported Breast Cancer Knowledge
Description: Measured pre-tool as 5-point Likert scale from "I know very little about breast cancer" (1) to "I know a lot about breast cancer" (5); analyzed as continuous variable.
Time Frame: Up to 1 hour
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Treatment Choice Reason
Description: Measured post-tool as an open text field.
Time Frame: Up to 1 hour
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Choice Confidence (Chambers et al., 2012)
Description: Measured post-tool as categorical 5-point Likert scale from "Not at all confident" (1) to "Very confident" (5); analyzed as continuous variable.
Time Frame: Up to 1 hour
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Information Needs Satisfaction (Adapted From Hess, 2012)
Description: Measured post-tool as 4-item scale, each item elicited on a 7-point Likert scale; items analyzed separately as continuous variables.
Time Frame: Up to 1 hour
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Knowledge Scale (De Novo)
Description: Measured post-tool (3 questions).
Time Frame: Up to 1 hour
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Knowledge Scale: Decision Quality Instrument (Adapted From Sepucha, et al., 2019)
Description: Measured post-tool (9 questions).
Time Frame: Up to 1 hour
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Preparation for Decision Making (PDMS) (Bennett, et al., 2010)
Description: Measured post-tool as 9-item scale, each item elicited on a 5-point Likert scale from "Not at all" (1) to "A great deal" (5); for each participant, the average score across 9 items is recorded and analyzed as a continuous variable.
Time Frame: Up to 1 hour
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Usability Question
Description: Measured post-tool as an open text field.
Time Frame: Up to 1 hour
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Aspects of Health Literacy Scale (AAHLS) (Chinn et al., 2013)
Description: Measured post-tool as a 7-item scale, each item elicited on a scale from "Rarely" (1) to "Often" (3).
Time Frame: Up to 1 hour
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Short Graph Literacy (Okan et al., 2019)
Description: Measured post-tool. Single score derived from 4 items, each scored as correct or incorrect. Correct answers are summed for a total "graph literacy score" (0-4).
Time Frame: Up to 1 hour
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Medical Maximizer Minimizer Scale (Scherer et al., 2020)
Description: Measured post-tool as categorical 6-point Likert scale from "I strongly lean toward waiting and seeing" (1) to "I strongly lean toward taking action" (6); analyzed as continuous variable.
Time Frame: Up to 1 hour
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Attitude Toward Risk (Zhang et al., 2019)
Description: Measured post-tool as an 8-item scale, each item elicited on a 5-point Likert scale from "Strongly disagree" (1) to "Strongly agree" (5).
Time Frame: Up to 1 hour
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Pain Tolerance (McCracken et al., 1992; Two Questions From Each Subscale)
Description: Measured post-tool as an 4-item scale, each item elicited on a 6-point Likert scale from "Never" (0) to "Always" (5).
Time Frame: Up to 1 hour
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Importance of Appearance (Borzekowski et al., 2000)
Description: Measured post-tool as a 4-item scale, each item elicited on a 6-point Likert scale from "Not at all important compared to other things in my life" (1) to "The very most important thing in my life" (6).
Time Frame: Up to 1 hour
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Cancer Fear (Lerman Worry Scale, 1991)
Description: Measured post-tool as a 3-item scale, each item elicited on a 5-point Likert scale from "Not at all" (1) to "Almost all the time" (5)
Time Frame: Up to 1 hour
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Current Health: Visual Analog Scale (Adapted From EQ-5D-3L, EuroQol Group, 1990)
Description: Self-reported health status (visual analog scale, 0-100).
Time Frame: Up to 1 hour
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Death, serious adverse events, and other (non-serious adverse events) were not assessed for the study.
Arm/Group | Standard Treatment Options + Active Monitoring | Standard Treatment Options
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-11-11): https://cdn.clinicaltrials.gov/large-docs/13/NCT03775213/Prot_001.pdf
  • Statistical Analysis Plan (2021-10-10): https://cdn.clinicaltrials.gov/large-docs/13/NCT03775213/SAP_002.pdf
  • Informed Consent Form (2021-08-02): https://cdn.clinicaltrials.gov/large-docs/13/NCT03775213/ICF_000.pdf